CLINICAL TRIAL: NCT00748553
Title: A Phase I/II Clinical Trial of the Hypomethylating Agent Azacitidine (Vidaza) With the Nanoparticle Albumin Bound Paclitaxel (Abraxane) in the Treatment of Patients With Advanced or Metastatic Solid Tumors and Breast Cancer
Brief Title: A Phase I/II Clinical Trial of Vidaza With Abraxane in Patients With Advanced/Metastatic Solid Tumors and Breast Cancer
Acronym: VA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI53993
Record Dates: First submitted 2008-09-04; First posted 2008-09-08 (Estimated); Results first posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-06

CONDITIONS: Advanced or Metastatic Solid Tumors; Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Azacitidine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Experimental): All participants enrolled.
  Interventions: Drug: Azacitidine (Vidaza); Drug: Nab-paclitaxel (Abraxane)

INTERVENTIONS:
Drug: Azacitidine (Vidaza) — 50mg/m2, 75mg/m2 or 100mg/m2 daily for 5 days for each 4-week cycle
  Other Names: Vidaza
Drug: Nab-paclitaxel (Abraxane) — 100mg/m2 weekly for 3 weeks of each 4-week cycle
  Other Names: Abraxane

SUMMARY:
The purpose of this clinical trial is to test whether treatment of patients with advanced or metastatic solid tumors or breast cancer with Abraxane plus Vidaza is safe and results in good tumor response. All patients enrolling in this study will receive treatment with Abraxane and Vidaza. Safety will be assessed by adverse events, laboratory results and performance status. Tumor response will be measured by RECIST criteria.

DETAILED DESCRIPTION:
The phase I part of the study will enroll patients with advanced or metastatic solid tumors who have failed at least one previous treatment. The purpose of the phase I part is to assess the safety of the investigational treatment and select the recommended phase II dose-regimen. The phase II part of the study will enroll patients with advanced or metastatic HER2-negative breast cancer who have not received treatment for their metastatic disease. The purpose of the phase II part of the study is to assess safety and efficacy of the investigational treatment in breast cancer. The study doctor will determine what phase patients will be enrolled in.

ELIGIBILITY:
Inclusion Criteria:

1. For phase I, any solid tumors, including lymphoma, that progressed or were stable as best response on at least one previous therapy and are evaluable.
2. For phase II, pathologically confirmed breast cancer, measurable disease, no prior treatments for recurrent or metastatic breast cancer.
3. Her-2/neu negative (Phase II)
4. Negative pregnancy test for female subjects
5. Women of childbearing potential should be advised to avoid becoming pregnant and men should be advised to not father a child while receiving treatment with azacitidine or nab-paclitaxel. investigator.
6. Male or female for phase I and female for phase II, >19 years of age and any race.

Exclusion Criteria:

1. Major surgery, radiotherapy, chemotherapy or investigational agents within 4 weeks of treatment day 1
2. Known brain metastases
3. Prior taxanes (except for adjuvant therapy more than 6 months prior to treatment day 1) (phase II)
4. Active infection requiring antibiotic therapy
5. History of allergy or hypersensitivity to nab-paclitaxel, albumin or a taxane
6. Grade 2 or greater motor or sensory neuropathy
7. Prior cytotoxic chemotherapy for recurrent or metastatic breast cancer (phase II portion)
8. Uncontrolled hypertension, arrhythmia, congestive heart failure or angina. Patients who have had a myocardial infarction or cardiac surgery should be at least 6 months from the event and free of active symptoms.
9. Known or suspected hypersensitivity to azacitidine or mannitol
10. Pregnant or breast feeding
11. Patients with advanced malignant hepatic tumors
12. Malignancy other than breast carcinoma (phase II)
13. Known HIV infection or chronic hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hung T Khong, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Azacitidine (Vidaza): 50mg/m2, 75mg/m2 or 100mg/m2 daily for 5 days for each 4-week cycle
  Nab-paclitaxel (Abraxane): 100mg/m2 weekly for 3 weeks of each 4-week cycle
- Phase II: Azacitidine is set at 75mg/m2 and Nab-paclitaxel is set at100mg/m2
Period: Overall Study
Arm/Group | Phase 1 | Phase II
Started | 16 | 14
Completed | 13 | 13
Not Completed | 3 | 1
Not completed — Adverse Event | 0 | 1
Not completed — disease progression | 2 | 0
Not completed — noncompliance | 1 | 0

BASELINE CHARACTERISTICS:
Population: In the Phase I cohort, two patients stopped during Cycle I due to disease progression, and one was removed in cycle 4 due to noncompliance. In the Phase II cohort, one patient opted out after 1 cycle because of toxicity.
Groups:
- Phase I: Azacitidine (Vidaza): 50mg/m2, 75mg/m2 or 100mg/m2 daily for 5 days for each 4-week cycle
  Nab-paclitaxel (Abraxane): 100mg/m2 weekly for 3 weeks of each 4-week cycle
- Total: Total of all reporting groups
Arm/Group | Phase II | Phase I | Total
Number analyzed (Participants) | 14 | 16 | 30
Age, Continuous [Median (Full Range); unit: years] | 65 [38 to 77] | 62 [21 to 83] | 63.5 [21 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 13 | 27
  Male | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 12 | 10 | 22
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 16 | 30

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Percentage of Participants Responding to Treatment
Description: Azacitidine is set at 75mg/m2 and Nab-paclitaxel is set at100mg/m2 based on the number of participants responding to treatment as measured per RECIST v1 criteria.
Time Frame: 6 months
Population: 16 patients were evaluable for toxicity. 13 were evaluable for response per RECIST v1.
Measure: Number (95% Confidence Interval); unit: percent of participants with response
Arm/Group | Phase 1
Number analyzed (Participants) | 13
percent of participants with response | 61.5 [35 to 87.95]

2. Primary Outcome: Phase II: Percentage of Participants With Objective Response Rate (ORR) Measured Using RECIST 1.0 Criteria
Description: Objective response rate (ORR) will be measured using RECIST 1.0 criteria. The best response, including complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD), for each patient will be summarized.
  For target lesions, Complete Response is defined as disappearance of all target lesions for at least 4 weeks; Partial Response consists of at least a 30% decrease in the sum of the LD of target lesions, taking as reference the baseline sum LD, for at least 4 weeks; Progressive Disease consists of at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions; Stable Disease consists of neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started.
Time Frame: 1.5 years
Population: Of the 14 patients enrolled on the Phase II portion of trial, one patient opted out off trial after 1 cycle because of toxicity.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II
Number analyzed (Participants) | 13
percentage of participants | 53.8 [26.7 to 80.9]

3. Secondary Outcome: Number of Participants With ER+ Status
Description: Tissue SPARC protein will be assessed using archival tumor blocks. In addition, in patients who have easily accessible tumors, such as lymph nodes, cutaneous or subcutaneous lesions, and who have consented to sample collection, biopsies will be taken twice: before cycle 1 day 1 treatment, and cycle 3 day 8 (+/- 3 days).
Time Frame: 2 years
Population: Of the 14 patients enrolled on the Phase II portion of trial, one patient opted out off trial after 1 cycle because of toxicity. Thirteen patients were evaluated for ER+ status.
Measure: Number; unit: participants were ER+
Arm/Group | Phase II
Number analyzed (Participants) | 13
participants were ER+ | 11

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PSF) is defined as the length of time during and after treatment in which a patient is living with a disease that does not get worse.
Time Frame: 2 years
Population: Data were not collected.
Arm/Group | Phase II
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Approximately 6 months. Adverse events will be assessed from the first day of treatment until at least 28 days after the last treatment or until all serious or study-related toxicities have resolved or are determined to be stable.
Description: Assessment of adverse events will include type, incidence, severity (graded by the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE], version3.0), timing, seriousness, and relatedness; and laboratory abnormalities.
  Baseline tumor-related signs and symptoms will be recorded as adverse events during the trial if they worsen in severity or increase in frequency.
Groups:
- Phase I and II: Azacitidine is set at 75mg/m2 and Nab-paclitaxel is set at100mg/m2
Arm/Group | Phase I and II
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 30/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I and II (N=30)
Alopecia (Skin and subcutaneous tissue disorders) | 10
Anemia (Blood and lymphatic system disorders) | 8
Anorexia (Metabolism and nutrition disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
chills (General disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Depression (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 6
Dizziness (Nervous system disorders) | 6
Dry mouth (Gastrointestinal disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 1
Edema (General disorders) | 4
Embolism (Vascular disorders) | 1
Fatigue (General disorders) | 18
Fever (General disorders) | 1
Headache (Nervous system disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hot flashes (Reproductive system and breast disorders) | 2
Hypoalbuminemia (Investigations) | 1
Injection Site Reaction (General disorders) | 1
Insomnia (Psychiatric disorders) | 2
White Blood Cell Decreased (Investigations) | 13
Memory impairment (Nervous system disorders) | 1
Mucositis (Gastrointestinal disorders) | 3
Muscle Weakness (Musculoskeletal and connective tissue disorders) | 5
Nail ridging (Skin and subcutaneous tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 11
Neuropathy (Nervous system disorders) | 14
Neutropenia (Investigations) | 11
Non-Cardiac chest pain (General disorders) | 1
Pain (General disorders) | 4
Sinusitis (Infections and infestations) | 1
Rash (Infections and infestations) | 4
Rhinitis (Infections and infestations) | 1
taste alteration (General disorders) | 5
Tremor (Nervous system disorders) | 1
Vomiting (Gastrointestinal disorders) | 7
Weight loss (Investigations) | 1
Dyspnea (Gastrointestinal disorders) | 1
Puritis (Skin and subcutaneous tissue disorders) | 2
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1
Weakness (General disorders) | 5
thrombocytopenia (Blood and lymphatic system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No